CLINICAL TRIAL: NCT04036474
Title: Development, Implementation, and Evaluation of School-based Smoking Prevention Education Program Among Non-smoking Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Esperanza Debby Ng, Research Assistant, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIUM/504/14/11/2/IREC650
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Smoking Behaviors
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking Prevention Education Program (Experimental): In addition to the lecture on the hazards of smoking, students received the SPEP intervention. The SPEP consisted of three lessons and each lesson took one to two hours to be implemented. The SPEP intervention was delivered to participants in their usual classroom setting, during school hours combined with relevant school subjects such as physical education class. The duration of SPEP intervention took approximately one month.
  Interventions: Other: Smoking Prevention Education Program
- Control (No Intervention): Immediately after the collection of baseline data, students received a one-time lecture on the hazards of smoking by the research assistant.

INTERVENTIONS:
Other: Smoking Prevention Education Program — The SPEP consisted of three lessons and each lesson took one to two hours to be implemented. SPEP was conducted through direct and indirect method. Direct method was conducted through lectures, question and answer, role play and educational videos. The tools used were video projectors and Power Point presentations. On the other hand, the indirect method was done through distributing of badge buttons and fridge magnets "Be Free from Smoking". This method brought a simple message to increase awareness among adolescents to prevent smoking uptake. All instruments and protocols in this intervention were pilot tested to confirm feasibility and cultural appropriateness.
  Arms: Smoking Prevention Education Program

SUMMARY:
Preventing smoking among adolescents is critical to end the epidemic of smoking in Malaysia. Despite the implementation of several smoking prevention programs, the prevalence of adolescent smoking and experimenting with tobacco in Malaysia is still increasing. Therefore, the purpose of this quasi-experimental study was to evaluate the effectiveness of Smoking Prevention Education Programs (SPEP) in preventing the smoking initiation among non-smoker adolescents based on their smoking status on follow-up and smoking intention, which includes; attitude, subjective norms, and perceived behavioural control as described by the Theory of Planned Behaviour. A total of 140 Primary five students (non- smokers) were involved in this study. Four schools in Kuantan district were randomly assigned to intervention and control groups. The intervention schools received a lecture on the hazards of smoking and SPEP intervention whereas the control schools received just a lecture on the hazards of smoking. The questionnaires and exhale carbon monoxide levels were first assessed at baseline and then again after three months.

ELIGIBILITY:
Inclusion Criteria:

* Primary school students (standard 5)
* 11years' old
* Non- smoker (CO level less than 4ppm) to maintain baseline never- smoker
* Both genders
* Consented by parent

Exclusion Criteria:

* Ex-smoker (self- reporting) and smoker (CO level more than 4ppm)
* Students unable to understand and read the national language (Bahasa Malaysia)
* Children with special needs

Ages: 11 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-01-28 (Actual); Study Completion 2017-01-28 (Actual)

PRIMARY OUTCOMES:
Number of students who smoke | 3 months
  Number of students who started smoking by the end of 3 months as assessed by a self-reported questionnaire and through measurement of exhaled CO levels using a handheld CO analyzer (piCO Smokerlyzer, Bedfont Scientific Ltd, England).

SECONDARY OUTCOMES:
Mean score of students' intention to smoke | 3 months
  Self-administering questionnaires were used to collect the baseline (before intervention) and follow-up (at 3 months post-intervention) data in this study. The questionnaires with translated versions (in English and Malay) were adapted and modified from the previous study by Melson (2014) based on the Theory of Planned Behaviour.
  Out of 24-items in the questionnaire, there are 3 items measuring behaviour intention on a 5-point Likert scale (1 = 'strongly disagree', 5 = 'strongly agree'), a higher value represents less intention to initiate smoking. Sample question for measuring behaviour intention include "I intend to be a non-smoker".
Mean score of students' attitudes towards smoking | 3 months
  Out of 24-items, there are 9 items measuring attitude on a 5-point Likert scale, a higher value represents an attitude of being in favor of smoking initiation. A sample question for measuring attitude include "I want to be a non-smoker".
Mean score of students' perception of subjective norms | 3months
  There are 6 items measuring subjective norms on the 5-point Likert scale, a higher value represents an individual experiencing social pressure not to initiate smoking. Sample question for measuring subjective norms include "Most people who are important to me think that I should be a non-smoker".
Mean score of students' perceived behavioural control | 3 months
  There are 6 items measuring perceived behaviour control on a 5-point Likert scale, a higher value represents an individual feeling in control from initiating smoking. Sample question for measuring perceived behavior control include "For me to be a non-smoker would be easy".

IPD SHARING:
Plan to Share IPD: No